CLINICAL TRIAL: NCT07114185
Title: A Prospective Study of Discomfort Symptoms in Patients With Aortic Disease After Endovascular Intervention
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT20250775B-R1
Record Dates: First submitted 2025-07-28; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Aortic Aneurysm and Dissection
Keywords: nursing; postoperative complication management
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients with aortic disease who received endovascular treatment

SUMMARY:
The incidence and severity of post-procedural discomfort were evaluated in patients undergoing endovascular repair for aortic disease across six symptom-related dimensions: immobilization-related issues, puncture site discomfort, adhesive-induced skin reactions, post-stent implantation syndrome, impairment in self-care ability, and physical/psychological stress responses.

DETAILED DESCRIPTION:
In this study, a customized postoperative discomfort symptom assessment questionnaire was developed based on patient-reported outcomes, aiming to systematically evaluate common discomfort symptoms experienced by patients with aortic disease after endovascular intervention. The questionnaire covers six core dimensions: immobilization-related discomfort, puncture site-related discomfort, adhesive-related skin reactions, post-stent implantation syndrome, decline in self-care ability, and psychosomatic stress responses. Each symptom within these dimensions was scored on a 0-4 scale according to severity: 0 indicates no symptoms; 1 indicates mild symptoms that are tolerable; 2 indicates moderate symptoms that affect daily life but are still tolerable; 3 indicates severe symptoms requiring medical intervention; and 4 indicates extremely severe symptoms that are intolerable and require emergency treatment.

Pain was evaluated using the Numeric Rating Scale (NRS). Skin reactions such as lesions, blisters, bruises, erythema, and rashes were quantified by measuring the longest and widest parts of the lesion using a flexible measuring tape. Self-care ability was assessed using the Activities of Daily Living (ADL) scale combined with patient self-evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with thoracoabdominal aortic disease
2. Patients who underwent endovascular treatment of the thoracoabdominal aorta via the femoral artery approach

Exclusion Criteria:

1. Aortic disease caused by infection
2. Aortic disease caused by trauma
3. Aortic disease treated by open abdominal surgery
4. Presence of systemic diseases uncontrollable by current medical standards (e.g., severe cardiac, pulmonary or hepatic dysfunction; advanced malignancy; cachexia; refractory severe coronary artery disease symptoms; coagulation disorders caused by genetic diseases, etc.)
5. Patients who have undergone endovascular aortic treatment via femoral artery access prior to this procedure due to other diseases (not related to the current aortic disease)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with aortic dissection undergoing endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative discomfort symptoms | 6, 24, and 48 hours postoperatively
  Based on six dimensions-immobilization-related, puncture site-related, adhesive-related skin reactions, aortic disease-related symptoms, self-care ability, and psychosomatic stress-patients were assessed at 6, 24, and 48 hours postoperatively using a structured questionnaire. The primary objective was to assess the incidence of postoperative complications and the severity of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol